CLINICAL TRIAL: NCT00748956
Title: Intranasal Administration of Neuropeptide Y in Healthy Male Volunteers
Acronym: NPY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dennis Charney (Other)
Responsible Party: Sponsor-Investigator, Dennis Charney, Dean, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GCO 05-0986; PT050986
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Mood Disorder; Anxiety Disorders
Keywords: Mood Disorder; Anxiety Disorders
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders | interventions — Neuropeptide Y

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose NPY (Experimental): Low dose, Receive 50 nmol dose of NPY
  Interventions: Drug: Low dose NPY
- High dose NPY (Experimental): High Dose, Receive 100 nmol dose of NPY
  Interventions: Drug: High dose NPY
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose NPY — 50nmol, administered intranasally
  Other Names: Neuropeptide Y
  Arms: Low dose NPY
Drug: High dose NPY — 100nmol administered intranasally
  Other Names: Neuropeptide Y
  Arms: High dose NPY
Drug: Placebo — placebo comparator (0nmol)) administered intranasally
  Arms: Placebo

SUMMARY:
There is growing evidence that neuropeptides act as neuronal messengers in the brain and have diverse functions that may include the regulation of mood and behavior. For example, neuropeptide Y (NPY) is thought to play a role in the adaptive stress response. The therapeutic application of neuropeptides for psychiatric disorders has been limited by difficult and unreliable penetration of the blood-brain barrier (BBB). However, recent data suggest that intranasal administration may provide a means of effectively delivering some of these neuropeptides to the brain. Thus far it is unclear if this is the case for NPY. The aims of this project are:

1. To evaluate, in 15 healthy male volunteers aged 25-45, the effect of intranasal NPY administration (0, 50 and 100 nmol) on its levels in cerebrospinal fluid (CSF), measured by means of lumbar puncture using an intraspinal catheter between L4 and L5, and in plasma, measured using an intravenous catheter in the forearm. One of the three treatments will be administered to each participant in a double-blind fashion. The 0 nmol condition will serve as the placebo control.
2. To test the effect of intranasal NPY administration on mood and anxiety.

DETAILED DESCRIPTION:
There is growing evidence that neuropeptides, including neuropeptide Y (NPY), act as neuronal messengers in the brain and have diverse neurobehavioral functions. Their therapeutic application for psychiatric disorders has been limited, however, by difficult and unreliable penetration of the blood-brain barrier (BBB). The BBB has prevented the use of many therapeutic agents for treating central nervous system (CNS) disorders. Several molecules have successfully been administered through intranasal delivery, however, thanks to the unique connection that the nerves involved in sensing odors and chemicals provide between the CNS and its environment.

NPY, the most abundant peptide in the mammalian brain, is co-localized with norepinephrine in sympathetic nerve fibers and has been of longstanding interest to our research group (Morgan et al., 2002; Morgan et al., 2003; Morgan et al., 2001; Morgan et al., 2000; Rasmusson et al., 2000; Rasmusson et al., 1998) because of its potential role in modulating mood and anxiety. NPY has been implicated as factor in the adaptive stress response (Thorsell et al., 1999), and has been shown to impact the consolidation of fear-related memories after shock (Flood et al., 1989). Clinically, lower plasma NPY levels have been correlated with greater psychological distress, increased symptoms of dissociation, and poorer performance among active duty military personnel. Acute stress in humans has been found to elicit NPY release, in a manner parallel to the changes in cortisol and norepinephrine that are usually seen, with a blunting of the plasma NPY response in response to yohimbine (Morgan et al., 2002). Baseline NPY levels in combat veterans with PTSD are reduced compared to healthy non-traumatized individuals (Rasmusson et al., 2000). Another study found that repeated exposure to traumatic stress, rather than the presence of PTSD or PTSD-type symptoms, is associated with a reduction in baseline plasma NPY (Morgan et al., 2003). A recent report found deceased CSF concentrations of NPY in patients with treatment resistant unipolar major depression (Heilig et al 2004). In summary, there has been suggestion from studies in patients with anxiety and mood disorders as well as healthy volunteers of an abnormal regulation of this peptide.

In this study, we will evaluate intranasal administration of NPY in healthy male volunteers ages 25-45 using a specialized delivery device. Pending the initial feasibility and tolerability in healthy volunteers, future protocols will examine the effect of intranasal NPY administration in patients with disorders such as PTSD, major depression, panic disorder, and social anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 25-45.
* No history of Axis I disorder as defined in the DSM-IV other than past nicotine abuse or dependence or adjustment disorder.

Exclusion Criteria:

* Nicotine or caffeine abuse or dependence within the preceding 3 months.
* History or complaint of nasal disorders or allergies.
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic.
* Significant obesity (BMI > 30), scoliosis, spinal stenosis or a history of lumbosacral laminectomy.
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG.
* Current use of any medications that have effects on CNS function.
* Prior sinonasal surgery, or significant nasal polyps as determined by nasal endoscopy.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Feder, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Dennis Charney, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Morgan CA 3rd, Rasmusson AM, Winters B, Hauger RL, Morgan J, Hazlett G, Southwick S. Trauma exposure rather than posttraumatic stress disorder is associated with reduced baseline plasma neuropeptide-Y levels. Biol Psychiatry. 2003 Nov 15;54(10):1087-91. doi: 10.1016/s0006-3223(03)00433-5. PMID 14625151
- [Background] Morgan CA 3rd, Wang S, Southwick SM, Rasmusson A, Hazlett G, Hauger RL, Charney DS. Plasma neuropeptide-Y concentrations in humans exposed to military survival training. Biol Psychiatry. 2000 May 15;47(10):902-9. doi: 10.1016/s0006-3223(99)00239-5. PMID 10807963
- [Background] Rasmusson AM, Hauger RL, Morgan CA, Bremner JD, Charney DS, Southwick SM. Low baseline and yohimbine-stimulated plasma neuropeptide Y (NPY) levels in combat-related PTSD. Biol Psychiatry. 2000 Mar 15;47(6):526-39. doi: 10.1016/s0006-3223(99)00185-7. PMID 10715359
- [Background] Rasmusson AM, Southwick SM, Hauger RL, Charney DS. Plasma neuropeptide Y (NPY) increases in humans in response to the alpha 2 antagonist yohimbine. Neuropsychopharmacology. 1998 Jul;19(1):95-8. doi: 10.1016/S0893-133X(97)00199-1. PMID 9608581
- [Background] Thorsell A, Carlsson K, Ekman R, Heilig M. Behavioral and endocrine adaptation, and up-regulation of NPY expression in rat amygdala following repeated restraint stress. Neuroreport. 1999 Sep 29;10(14):3003-7. doi: 10.1097/00001756-199909290-00024. PMID 10549813
- [Background] Flood JF, Baker ML, Hernandez EN, Morley JE. Modulation of memory processing by neuropeptide Y varies with brain injection site. Brain Res. 1989 Nov 27;503(1):73-82. doi: 10.1016/0006-8993(89)91706-x. PMID 2611661
- [Background] Heilig M. The NPY system in stress, anxiety and depression. Neuropeptides. 2004 Aug;38(4):213-24. doi: 10.1016/j.npep.2004.05.002. PMID 15337373
- [Background] Eaton K, Sallee FR, Sah R. Relevance of neuropeptide Y (NPY) in psychiatry. Curr Top Med Chem. 2007;7(17):1645-59. doi: 10.2174/156802607782341037. PMID 17979774
- [Background] Nikisch G, Agren H, Eap CB, Czernik A, Baumann P, Mathe AA. Neuropeptide Y and corticotropin-releasing hormone in CSF mark response to antidepressive treatment with citalopram. Int J Neuropsychopharmacol. 2005 Sep;8(3):403-10. doi: 10.1017/S1461145705005158. Epub 2005 Mar 23. PMID 15784158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Started | 0 | 5 | 5
Completed | 0 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose NPY | High Dose NPY | Placebo | Total
Number analyzed (Participants) | 0 | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0
  Between 18 and 65 years |  | 5 | 5 | 10
  >=65 years |  | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0 | 0
  Male |  | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Levels of NPY in CSF
Description: Levels of Neuropeptide Y in the cerebrospinal fluid
Time Frame: on study day 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Number analyzed (Participants) | 0 | 5 | 5
pg/mL |  | 329.4 (119.9) | 351.0 (41.6)

2. Secondary Outcome: Systematic Assessment of Treatment-Emergent Effects (SAFTEE)
Description: Number of participants with serious adverse events
Time Frame: on study day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Number analyzed (Participants) | 0 | 5 | 5
Participants | 0 | 0 | 0

3. Secondary Outcome: Appetite Scale
Description: measure in 2 hours post intranasal administration
Time Frame: on study day 2
Population: data not collected
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Post-sleep Questionnaire
Description: measure in the morning
Time Frame: on study day 2
Population: data not collected
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Quick Inventory of Depressive Symptoms (QIDS)
Description: measure in 2 hours post intranasal administration
Time Frame: on study day 2
Population: data not collected
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Profile of Mood States (POMS)
Description: measure in 2 hours post intranasal administration and on the next morning
Time Frame: on study day 2
Population: data not collected
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Low Dose NPY | High Dose NPY | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/5 | 1/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose NPY (N=0) | High Dose NPY (N=5) | Placebo (N=5)
Headache and Nausea (Nervous system disorders) | 0 | 0 | 1 — ER evaluation for headache and nausea
Headache (Nervous system disorders) | 0 | 1 | 0 — Headache requiring hospitalization

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes